CLINICAL TRIAL: NCT03980691
Title: Effect of Chidamide Combined With CAT-T or TCR-T Cell Therapy on HIV-1 Latent Reservoir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou 8th People's Hospital (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Linghua LI, Vice Chief physician, Guangzhou 8th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20171126V1
Record Dates: First submitted 2019-06-07; First posted 2019-06-10 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: HIV/AIDS
Keywords: Chidamide,CAR cell therapy,TCR cell therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Intervention Model Description: The control arm includes HIV-infected patients without receiving cellar therapy combined with Chidamide whose HIV-1 has been successfully suppressed after cART.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chidamide combined with CAR-T or TCR-T cell therapy (Experimental): Receiving chidamide combined with CAR-T or TCR-T cell therapy based on based on cART after attaining plasma HIV suppression (plasma HIV RNA <50 cp/ ml) and CD4+ cell count more than 350 cells/ul over 1 year by cART without active HCV or HBV infection or opportunistic infections.
  Interventions: Biological: Chidamide with CAR-T or TCR-T cell therapy
- without intervention (No Intervention): Not receiving chidamide combined with CAR-T or TCR-T cell therapy but continuing cART after attaining plasma HIV suppression (plasma HIV RNA <50 cp/ml) and CD4+ cell count more than 350 cells/ul over 1 year by cART, without active HCV or HBV infection or opportunistic infections.

INTERVENTIONS:
Biological: Chidamide with CAR-T or TCR-T cell therapy — HIV-1 specific therapy
  Arms: Chidamide combined with CAR-T or TCR-T cell therapy

SUMMARY:
To study the safety and effectiveness of the combination of Chidamide with Chimeric Antigen Receptor(CAR)-T or T cell receptor(TCR)-T cell therapy on HIV patients based on cART.

DETAILED DESCRIPTION:
Despite the advent of combined antiretroviral therapy (cART), the persistence of viral reservoirs remains a major barrier to cure human immunodeficiency virus type 1 (HIV-1) infection. Recently, the shock and kill strategy, by which such reservoirs are eradicated following reactivation of latent HIV-1 by latency-reversing agents (LRAs), has been extensively practiced. It is important to reestablish virus-specific and reliable immune surveillance to eradicate the reactivated virus-harboring cells. Some studies have shown that Chidamide can highly activate the HIV reservoirs. The VC-CAR-T cells effectively induced the cytolysis of LRA-reactivated HIV-1-infected CD4 T lymphocytes isolated from infected individuals receiving suppressive cART. Our previous study demonstrated that the special features of genetically engineered CAR-T cells make them a particularly suitable candidate for therapeutic application in efforts to reach a functional HIV cure. The purpose of this study is to evaluate the safety and efficacy of Chidamide together with Chimeric Antigen Receptor(CAR)-T or T cell receptor(TCR)-T cell therapy based on cART in HIV-infected adults whose plasma HIV has been successfully suppressed after cART.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection confirmed
2. Receiving cART more than 12 months.
3. HIV viral-load < 50 copies/ml and CD4 cell count more than 350 cells/ul.
4. Without serious liver , heart, liver and kidney diseases.
5. The subjects know about the study and volunteer to attend the research and sign the informed consent.

Exclusion Criteria:

1. With active HBV or HCV infection, or serious opportunistic infections.
2. With serious chronic disease such like diabetes, the mental illness,et al
3. History of suffering from pancreatitis during cART .
4. Pregnant or breast-fed.
5. With poor adherence.
6. Unable to complete follow up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-associated adverse events | 6 Months
  To observe the adverse events of intervention n HIV-infected patients during the study.

SECONDARY OUTCOMES:
HIV reservoir | 6 Months
  To assay the HIV loads in the peripheral blood Mono-nuclear cells and plasma

OTHER OUTCOMES:
HIV-specific immunity | 6 Months
  The number of HIV-specific CD4,CD8,VC-CAR-T and TCR-T cells after receiving the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Cai, Bachelor, Principal Investigator — Guangzhou 8th People's Hospital China, Guangdong
Locations (1):
- Guangzhou 8th People's Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Dotti G, Gottschalk S, Savoldo B, Brenner MK. Design and development of therapies using chimeric antigen receptor-expressing T cells. Immunol Rev. 2014 Jan;257(1):107-26. doi: 10.1111/imr.12131. PMID 24329793
- [Background] Liu C, Ma X, Liu B, Chen C, Zhang H. HIV-1 functional cure: will the dream come true? BMC Med. 2015 Nov 20;13:284. doi: 10.1186/s12916-015-0517-y. PMID 26588898
- [Background] Kuai Q, Lu X, Qiao Z, Wang R, Wang Y, Ye S, He M, Wang Y, Zhang T, Wu H, Ren S, Yu Q. Histone deacetylase inhibitor chidamide promotes reactivation of latent human immunodeficiency virus by introducing histone acetylation. J Med Virol. 2018 Sep;90(9):1478-1485. doi: 10.1002/jmv.25207. Epub 2018 May 25. PMID 29704439
- [Background] Yang W, Sun Z, Hua C, Wang Q, Xu W, Deng Q, Pan Y, Lu L, Jiang S. Chidamide, a histone deacetylase inhibitor-based anticancer drug, effectively reactivates latent HIV-1 provirus. Microbes Infect. 2018 Oct-Nov;20(9-10):626-634. doi: 10.1016/j.micinf.2017.10.003. Epub 2017 Nov 8. PMID 29126877
- [Background] Kobayashi Y, Gelinas C, Dougherty JP. Histone deacetylase inhibitors containing a benzamide functional group and a pyridyl cap are preferentially effective human immunodeficiency virus-1 latency-reversing agents in primary resting CD4+ T cells. J Gen Virol. 2017 Apr;98(4):799-809. doi: 10.1099/jgv.0.000716. Epub 2017 Apr 27. PMID 28113052
- [Result] Liu B, Zou F, Lu L, Chen C, He D, Zhang X, Tang X, Liu C, Li L, Zhang H. Chimeric Antigen Receptor T Cells Guided by the Single-Chain Fv of a Broadly Neutralizing Antibody Specifically and Effectively Eradicate Virus Reactivated from Latency in CD4+ T Lymphocytes Isolated from HIV-1-Infected Individuals Receiving Suppressive Combined Antiretroviral Therapy. J Virol. 2016 Oct 14;90(21):9712-9724. doi: 10.1128/JVI.00852-16. Print 2016 Nov 1. PMID 27535056